CLINICAL TRIAL: NCT02821559
Title: Biweekly Versus Triweekly Raltitrexed With Oxaliplatin (With or Without Bevacizumab) in First-line Metastatic Colorectal Cancer
Acronym: EROS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EROS; 2011-005811-96 (EudraCT Number)
Record Dates: First submitted 2016-03-29; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; raltitrexed; oxaliplatin; bevacizumab; biweekly; triweekly
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

ARMS (2):
- triweekly then biweekly (Experimental): The arm A consisted of 2 cycles of triweekly TOMOX (standard dose 3mg/m2 of Raltitrexed in 15-minutes infusion, and 130mg/m2 of oxaliplatin in 2h infusion, every 3 weeks), followed by 2 cycles of biweekly TOMOX (2mg/m2 of Raltitrexed in 15-minutes infusion, and 85mg/m2 of oxaliplatin in 2h infusion, every 2 weeks).
  Interventions: Drug: TOMOX; Drug: Bevacizumab
- biweekly then triweekly (Experimental): The arm B consisted of the reserve sequence starting with 2 cycles of biweekly TOMOX followed by 2 cycles of triweekly TOMOX regimen.
  Interventions: Drug: TOMOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: TOMOX
  Other Names: Tomudex-Oxaliplatin; Raltitrexed-Oxaliplatin
Drug: Bevacizumab — Bevacizumab was allowed and used at 7,5 mg/kg or 5 mg/kg every 2 weeks.

SUMMARY:
Raltitrexed is a potent thymidylate synthase (TS) inhibitor. Conversely to 5-fluorouracil (5FU), raltitrexed can be administered safely in patients with cardiovascular disease, as well as in patients with dihydropyrimidine dehydrogenase deficit. Since raltitrexed is administered in 15-minutes infusion, complications related to continuous infusion can be avoided, and it becomes a potential good candidate for locoregional treatments as hepatic intra-arterial or intra-peritoneal infusion. Despite these potential benefits over 5FU, clinical trials failed in their temptation to replace the 5FU in colorectal cancer patients, mainly due to raltitrexed toxicity at 3mg/m2 every 3 weeks. Oxaliplatin has demonstrated a synergic effect when combined with TS inhibitors, and its association with raltitrexed was evaluated at 130mg/m2 of oxaliplatin and 3mg/m2 of raltitrexed, every 3 weeks. Actually, one of the first-line standard regimens in metastatic colorectal cancer patients is the biweekly FOLFOX (85mg/m2 of oxaliplatin, and infusional 5FU) plus bevacizumab regimen, since a significant progression-free survival (PFS) benefit was observed over FOLFOX plus placebo. Biweekly administration of raltitrexed at 2mg/m2 demonstrated a favorable toxicity profile even in patients aged >65 years. Besides, the association of raltitrexed, oxaliplatin and bevacizumab seems safe.

Then, the investigators decided to perform a randomized pharmacokinetic comparative study between biweekly TOMOX (raltitrexed 2 mg/m2 and oxaliplatin 85mg/m2) and triweekly TOMOX (raltitrexed 3 mg/m2 and oxaliplatin 130mg/m2) regimens in metastatic colorectal cancer patients, in a "ping-pong" crossover strategy to reduce the intra-individual variability. Bevacizumab was allowed at the dose of 5mg/kg or 7.5mg/kg, in biweekly and triweekly schedules, respectively. The secondary end-points were, objective response rate evaluated by RECIST 1.1 criteria, PFS, overall survival (OS), toxicity, and the comparison of toxicity between two arms for the first 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* performance status (ECOG-PS) of 0 or 1
* patient with histologically proven colorectal cancer with distant metastases
* measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* life expectancy > 12 months
* signed written informed consent

Exclusion Criteria:

* prior chemotherapy at metastatic stage
* presence of brain or meningeal metastases
* other malignancies in the past 5 years with the exception of adequately treated carcinoma in situ of the cervix and squamous or basal cell carcinoma of the skin
* preexisting peripheral neuropathy
* known hypersensitivity to any component of the study treatment
* any psychiatric condition compromising the understanding of information or conduct of the study
* pregnancy, breast-feeding or absence of adequate contraception for fertile patients
* patient under guardianship, curator or under the protection of justice

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evolution of Raltitrexed plasma levels | at 5 minutes, at 40 minutes, at 2 hours, at 7,5 hours, at 24 hours and at 14 days after each raltitrexed administration
  pharmacokinetic study

SECONDARY OUTCOMES:
treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  comparison of number of treatment-related adverse events between two arms
objective response rate evaluated by RECIST 1.1 criteria | 3 months
progression-free survival (PFS) | through study completion, an average of 2 years
  from date to randomization to date of first progression of the disease
overall survival (OS) | through study completion, an average of 2 years
  from date to randomization to date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Besançon, Besançon, France